CLINICAL TRIAL: NCT05304871
Title: A Randomized, Double Blind, Placebo-controlled Clinical Trial Assessing the Utility of Antibiotic Prophylaxis Prior to Totally Implanted Venous Access Device (TIVAD) Insertion
Brief Title: Randomized Assessment of Antibiotic Prophylaxis Prior to Port Placement
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Eric K. Hoffer, Director, Vascular and Interventional Radiology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY02000371
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Vascular Access Ports
MeSH Terms: interventions — Cefazolin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo and antibiotic packaged similarly, code identified by Investigational Pharmacy. Patients and providers will not know which had been administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): patients receive saline infusion prior to port placement
  Interventions: Other: saline
- antibiotic (Experimental): patients receive antibiotic (Cefazolin 2 g) infusion prior to port placement
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin — infusion
  Arms: antibiotic
Other: saline — infusion
  Other Names: placebo
  Arms: placebo

SUMMARY:
A randomized, double blind, placebo-controlled clinical trial assessing the utility of antibiotic prophylaxis prior to Totally Implanted Venous Access Device (TIVAD) insertion.

DETAILED DESCRIPTION:
To assess the effectiveness of peri-procedural antibiotic prophylaxis in the reduction of TIVAD placement-related infection, study will compare placebo (normal saline (0.9% NaCl)) 50 cc IV 1:1 to the standard clinical antibiotic prophylaxis dose. The primary endpoint is cumulative incidence of local TIVAD surgical site infection (as determined by the CDC criteria for a deep and/or superficial SSI) or a central line associated blood stream infection at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring TIVAD insertion for long-term central venous access
* Patients able to give informed consent to participate in the study.

Exclusion Criteria:

* taking long-term antibiotics
* unable to give consent to participate in the study
* Patients that have a known infection at time of the procedure (as documented in e-DH).
* Patients with a planned surgical procedure within 30 days of initial TIVAD insertion.
* Patients that are currently on antibiotics or have received antibiotics within the last week.
* Patients with allergies to cefazolin.
* Patients with an absolute neutrophil count of less than 500/mm3
* Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with surgical site infection | 30 days after procedure
  surgical site infection; Effectiveness will be evaluated by comparing infection rates between patients that receive systemic prophylactic antibiotic and those that receive a placebo
Number of participants with CRBSI | 30 days after procedure
  catheter-related bloodstream infection (CRBSI); Effectiveness will be evaluated by comparing infection rates between patients that receive systemic prophylactic antibiotic and those that receive a placebo

SECONDARY OUTCOMES:
Average cost of systemic prophylactic antibiotic administration compared to the cost of treating TIVAD insertion related infections | 30 days after procedure
  expense associated with catheter or catheter-related complication care; compare the costs of systemic prophylactic antibiotic administration, prior to totally implanted central venous access device (TIVAD) insertion, to the cost of treating TIVAD insertion related infections

IPD SHARING:
Plan to Share IPD: No